CLINICAL TRIAL: NCT06737289
Title: PRECISION OF SURGICAL GUIDES FOR PLACEMENT OF EXTRA-LARGE DENTAL IMPLANTS. A PILOT STUDY
Brief Title: SURGICAL GUIDES EFFECTIVENESS
Acronym: ASG-EI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Jesús Torres García Denche, Associate Profesor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.I. 24/728-E
Record Dates: First submitted 2024-11-30; First posted 2024-12-17 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Atrophic Maxilla
MeSH Terms: conditions — Atrophic Maxilla

STUDY DESIGN:
Intervention Model Description: Split Mouth Design
Who Masked: Participant, Outcomes Assessor
Masking Description: blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guide Surgery Arm (Experimental): Use of Surgical Guide
  Interventions: Procedure: Surgical Guide
- Control (Placebo Comparator): Hand Free Implant Placement
  Interventions: Procedure: Surgical Guide

INTERVENTIONS:
Procedure: Surgical Guide — Placing extralarge implats for rahabilitation atrophic maxilla

SUMMARY:
The use of zygomatic implants is a technique that is becoming more and more widespread in daily clinical practice, however, few professionals feel safe and confident in performing this type of procedure. We therefore believe that a line of research focused on simplifying this technique will have an extraordinary impact on the safety of both patients and surgeons. Currently, new surgical guides have emerged that guarantee greater precision in the placement of zygomatic implants. However, no comparative clinical studies have yet been performed to evaluate the degree of accuracy of guided implant placement compared to the conventional freehand technique.

DETAILED DESCRIPTION:
The primary objective of the study is to study the accuracy of the use of guided surgical splints compared to traditional freehand zygomatic implant placement.

The secondary objectives are:

* To compare the magnitude of variations depending on implant length by superimposing postoperative CT scans using 3DSlicer® (http://www.slicer.org) and exocad® software.
* To compare the magnitude of the variations depending on the location of the implant by superimposing postoperative and postoperative CT scans using 3DSlicer® (http://www.slicer.org) and exocad® software.
* To assess the clinical relevance of cogomatic implant placement using guided surgical splinting on pain parameters and surgical time.

ELIGIBILITY:
Inclusion Criteria:

• Age between 18-80 years of age, patients who sign the informed consent form and patients who consent to undergo preoperative and postoperative orthopantomography and CT scans.

Exclusion Criteria:

* Smoking (more than 10 cigarettes per day).
* Alcoholism (more than 25g/day in women and more than 40g/day in men according to WHO criteria),
* Oncological treatment (history of treatment in the last 6 months or current treatment with chemotherapy or radiotherapy).
* History of head and neck radiotherapy.
* Allergic to anesthetics or antibiotics.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-06-12 (Estimated); Study Completion 2025-10-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Surgical Guides in implant placement | 12 months
  Accuracy of Surgical Guides in terms of Radiological differences in implant placement. The primary outcome is to measure the differences existing between implant planificación and final implant placement. First, a computed tomography (CT) scan will be performed to plan the placement of the zygomatic implants. Once the implants have been placed in both groups, another CT scan will be performed to evaluate the following parameters using 3DSlicer® software (http://www.slicer.org). Three-dimensional lateral apical implant deviation and three-dimensional lateral neck implant deviation respect to the original digital planning will be evaluated by superimposing images.
  3D lateral deviations will be measured in mm in relation with original planning.
  Also deviations in degrees between the original planning and the final placements will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: JEsus Torres, PhD, Principal Investigator — UCM
Locations (2):
- Spain (2):
  - Jesus, Madrid
  - UCM, Madrid